CLINICAL TRIAL: NCT04962724
Title: A Phase 1, Open-label, 2-part, Single-dose Study of the Absorption, Metabolism, and Excretion of Oral [14C]-Xevinapant, and Absolute Oral Bioavailability of Xevinapant in Healthy Male Subjects
Brief Title: A Study to Evaluate the Absorption, Metabolism, and Excretion and Absolute Bioavailability of Xevinapant in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Debiopharm International SA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Debio 1143-108
Record Dates: First submitted 2021-06-21; First posted 2021-07-15 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers
Keywords: Xevinapant; Absorption, Distribution, Metabolism and Excretion (ADME); Mass balance; Absolute bioavailability
MeSH Terms: interventions — Solutions; Infusions, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Radiolabeled Xevinapant Oral Solution (Experimental): Participants will receive:
  • single oral dose of [14C]-xevinapant, as an oral solution
  Interventions: Drug: Radiolabelled Xevinapant 200 mg (Oral Solution)
- Radiolabeled Xevinapant Intravenous Solution + Xevinapant Oral Solution (Experimental): Participants will receive:
  • single oral dose of xevinapant, as an oral solution followed by an IV bolus of [14C]-xevinapant, solution for infusion
  Interventions: Drug: Radiolabelled Xevinapant 100 μg (IV Solution); Drug: Xevinapant 200 mg (Oral Solution)

INTERVENTIONS:
Drug: Radiolabelled Xevinapant 200 mg (Oral Solution) — [14C]-Xevinapant 200 mg administered as an oral solution on Day 1 of Part 1, containing approximately 100 microcurie (μCi) [3.7 megabecquerel (MBq)] in fasted conditions.
  Arms: Radiolabeled Xevinapant Oral Solution
Drug: Radiolabelled Xevinapant 100 μg (IV Solution) — 100 μg [14C]-xevinapant single dose administered as an IV bolus on Day 1, containing approximately 0.2 μCi [7.4 kilobecquerel (kBq)].
  Arms: Radiolabeled Xevinapant Intravenous Solution + Xevinapant Oral Solution
Drug: Xevinapant 200 mg (Oral Solution) — Xevinapant 200 mg administered as an oral solution on Day 1 of Part 2 in fasted conditions
  Arms: Radiolabeled Xevinapant Intravenous Solution + Xevinapant Oral Solution

SUMMARY:
The purpose of the study is to determine absorption, metabolism, and excretion of a single oral dose of [14C]-xevinapant. This information will enable assessment of absorption and clearance mechanisms of [14C]-xevinapant as well as identify metabolites. In addition, the study will allow to determine absolute bioavailability of xevinapant and understand its intravenous pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: Males of any race, between 35 and 65 years of age, inclusive. Part 2: Males of any race, between 18 and 65 years of age, inclusive
* Body mass index between 18.0 and 30.0 kilograms per meter square (kg/m^2), inclusive
* Weight between 50 kilograms (kg) and 110 kg, inclusive
* History of a minimum of 1 bowel movement per day.
* Willing to adhere to the prohibitions and restrictions specified in the study protocol

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee)
* History of alcohol consumption of >21 units per week. One unit of alcohol equals 12 ounce (oz) [360 millilitre (mL)] beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine.
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 90 days prior to dosing, or less than 5 times the half-life, whichever is longer, prior to administration of study drug
* Poor peripheral venous access
* Have participated in any clinical study involving a radiolabeled investigational product within 12 months prior to check-in.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Mass Balance Recovery Measured Through Total Radioactivity Excreted in Expired Air, Urine and Feces | Up to Day 29
Area Under Concentration-Time Curve From Time Zero to Infinity (AUC0-infinity); Time 0 to 24 Hours (AUC0-24); Time 0 to Last Quantifiable Concentration (AUC0-last) of Total Radioactivity in Blood and Plasma, and of Xevinapant and Metabolite in Plasma | Up to Day 29
Maximum Observed Concentration (Cmax) of Total Radioactivity in Blood and Plasma, and of Xevinapant and Metabolite in Plasma | Up to Day 29
Time to Maximum Observed Concentration (Tmax) of Total Radioactivity in Blood and Plasma, and of Xevinapant and Metabolite in Plasma | Up to Day 29
Apparent Terminal Elimination Half-life (T1/2) of Total Radioactivity in Blood and Plasma, and of Xevinapant and Metabolite in Plasma | Up to Day 29
Apparent Volume of Distribution During Terminal Phase (Vz/F) of Total Radioactivity in Blood and Plasma, and of Xevinapant and Metabolite in Plasma | Up to Day 29
Apparent Total Clearance (CL/F) of Total Radioactivity in Blood and Plasma and of Xevinapant and Metabolite in Plasma | Up to Day 29
Renal Clearance (CLr) of Total Radioactivity, Xevinapant and Metabolite | Up to Day 29
Xevinapant Metabolite Concentrations in Urine, Feces, Blood and Plasma | Up to Day 8
Absolute Bioavailability (F) of Xevinapant in Plasma | Up to Day 5
  Absolute Bioavailability (F) = (AUC0-infinity [oral]/ dose [oral]) /(AUC0-infinity [IV]/ dose [IV])

SECONDARY OUTCOMES:
Blood to Plasma Ratio of Xevinapant and Metabolite | Up to Day 8
Plasma Protein Binding Expressed as Fraction unbound, fu of Xevinapant | Up to Day 8
Safety and Tolerability as Measured by Number of Participants With Treatment-Emergent Adverse Events | Up to Day 29
Safety and Tolerability as Measured by Number of Participants With Clinically significant Laboratory Abnormalities | Up to Day 29
Safety and Tolerability as Measured by Number of Participants With Clinically significant 12-lead ECG Parameters Abnormalities | Up to Day 29
Safety and Tolerability as Measured by Number of Participants With Clinically significant Vital Signs Abnormalities | Up to Day 29
Safety and Tolerability as Measured by Number of Participants With Clinically significant Physical Examination Abnormalities | Up to Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Labcorp Clinical Research Unit, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided